CLINICAL TRIAL: NCT03624985
Title: The Effect of Perioperative Intravenous Lidocaine Infusion on Opioid Consumption After Lumbar Spine Surgery
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Subjects had a high dropout rate. Of 61 consented, 24 did not participate. Reasons: Surgical cancellations; changing procedure type after consent; and staffing issues. The dropout rate of 39% was considered a barrier to publication.
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Tim Dominick, Anesthesiologist, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHRMS 18-0111
Record Dates: First submitted 2018-06-13; First posted 2018-08-10 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative; Opioid Use
Keywords: lidocaine; lumbar spine surgery; postoperative pain; opioid reduction
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized, controlled, double-blind study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous Lidocaine Infusion (Experimental): Patients will be randomly assigned to receive 1 mg/kg lidocaine bolus and intraoperative infusion of 2 mg/min.
  Interventions: Drug: Intravenous Lidocaine Infusion
- Placebo Infusion (Placebo Comparator): Patients will be randomly assigned to receive a 1mg/kg bolus of water with 5% dextrose and an intraoperative infusion of 2mg/min. of water with 5% dextrose.
  Interventions: Drug: Placebo Infusion

INTERVENTIONS:
Drug: Intravenous Lidocaine Infusion — Patients will be randomly assigned to receive 1 mg/kg lidocaine bolus and intraoperative infusion of 2 mg/min.
  Other Names: IV Lidocaine Infusion
  Arms: Intravenous Lidocaine Infusion
Drug: Placebo Infusion — Patients will be randomly assigned to receive a 1mg/kg bolus of water with 5% dextrose and an intraoperative infusion of 2mg/min. of water with 5% dextrose
  Other Names: Placebo; Control; Comparator
  Arms: Placebo Infusion

SUMMARY:
The purpose of this study is to determine whether an infusion of lidocaine during surgery can reduce the need for postoperative opioid pain medication use in patients undergoing lumbar spine surgery.

Participants will be recruited by spine surgeons from their pool of patients who are presenting for surgery at University of Vermont Medical Center. If they agree to participate, patients will be assigned at random to receive either an infusion of lidocaine during surgery, or an infusion of saline with 5% dextrose. Subjects will also be asked to complete a 15-item questionnaire that asks about health, quality of life, and level of pain, at three timepoints. Patients will also be asked to rate their level of pain at multiple timepoints after surgery, and we will collect the additionally data from patients' medical records.

DETAILED DESCRIPTION:
Lidocaine has analgesic and anti-inflammatory effects. It has been shown to reduce early postoperative pain and nausea. Additionally, lidocaine has been shown to have positive effects in the recovery of bowel function, with a reduction in time to first flatus, first bowel sounds, first bowel movement, and is associated with a reduction of ileus. Because of these facts, lidocaine infusion has become part of enhanced recovery pathways after bowel surgery at our institution and others.

There are few trials examining the use of lidocaine for orthopedic procedures and many of these studies have contradictory adults. An article by Martin et al. found no benefit in pain or recovery after total hip arthroplasty. By contrast, Farag and colleagues found that lidocaine significantly improves postoperative pain after major spine surgery. Additionally, quality of life scores at one and three months after surgery were significantly higher in the lidocaine group. When our Spine Surgery Analgesic Protocol for major spine surgery at University of Vermont Medical Center was revised in 2015, a lidocaine infusion was added to the protocol.

Studies for lidocaine use in minor lumbar surgery are scant. In one study of 50 patients in Korea, patient pain scores and fentanyl consumption were significantly lower in the lidocaine infusion group (1.5 mg/kg bolus plus 2 mg/kg/hr infusion) at 2, 4, 8, 12 and 24 hours after surgery. Of note, the Cleveland Clinic Outcomes group is currently enrolling 440 patients in a study in which half will receive lidocaine and ketamine infusions.

A reduction in opioid use may lead to the potential reduction of opioid-related side effects, such as nausea, constipation, and hyperalgesia, as well as more serious consequences such as respiratory depression and abuse. There is also the possibility of a length of stay reduction which has potential financial benefits.

This is a randomized, controlled, double-blind study involving patients undergoing one- or two-level posterior lumbar instrumented spinal fusion with or without decompression.

The University of Vermont Medical Center operating rooms will be utilized for this investigation. For the study group, we plan to prospectively recruit 140 patients 18-75 years of age. Recruitment will be done by the participating orthopedists and neurosurgeons, from their own patients. After an informed consent discussion, patients will be randomly assigned to receive 1 mg/kg lidocaine bolus and intraoperative infusion of 2 mg/min (intervention arm) or no lidocaine (control arm). All patients will receive adequate pain control medication according to their needs. Subjects will complete the 15-question Quality of Recovery assessment at baseline and at 36 and 60 hours after surgery. Using the electronic medical system, the following information with extracted: Total morphine equivalent used in house at 36 hours, total morphine equivalents used at 60 hours, visual analog scale pain scores at 4, 8, 12, 24, 36, and 60 hours, length of stay, incidence of nausea requiring medication, time to first flatus, and time to first bowel movement. Subjects will receive a patient-controlled analgesia pump for the first 36 hours after surgery.

Randomization will be performed by the University of Vermont Medical Center Investigational Pharmacy Drug Service (IDS). IDS will generate a table of random numbers and assign those numbers in a 1:1 ratio of active drug to placebo, in blocks of 4. Following informed consent, a member of the study team will notify IDS, which will prepare syringes for the bolus dose and a bag for the infusion, both containing either active drug or placebo. The syringes and bag will be labeled with the subject's name, medical record number, and randomization number.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing one- or two-level posterior lumbar fusion with or without decompression at University of Vermont Medical Center
* 18-75 years of age
* Signed consent form

Exclusion Criteria:

* Allergy to lidocaine
* Contraindication to lidocaine, such as substantial hepatic impairment (alanine aminotransferase or aspartate transaminase more than twice normal), renal impairment (serum creatinine >2 mg/dl)
* Seizures or a history of seizure disorder
* Congestive heart failure
* Arrythmias
* Chronic opioid use >45 mg morphine equivalent per day
* Trauma patients
* Inter-body fusions
* Severe psychiatric comorbidities
* Planned epidural anesthesia or analgesia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-10-14 (Actual); Study Completion 2019-10-14 (Actual)

PRIMARY OUTCOMES:
Total morphine equivalent consumed at 24 hours after surgery | 24 hours postoperatively
  Subjects will receive a patient-controlled analgesia pump for the first 24 hours after surgery. Total morphine equivalent will be calculated according to the Centers for Disease Control and Prevention conversion factor for calculating morphine milligram equivalents.

SECONDARY OUTCOMES:
Total morphine equivalent consumed at 48 hours after surgery | 48 hours postoperatively
  Electronic medical records will be reviewed to total opioids received after the patient-controlled analgesia pump is discontinued. Total morphine equivalent will be calculated according to the Centers for Disease Control and Prevention conversion factor for calculating morphine milligram equivalents.
Pain score 4 hours post-operation | 4 hours postoperatively
  Visual analog scale pain scores 4 hours after the end of the operation.
  The visual analog scale is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The patient marks a point on the line that matches the amount of pain they feel.
  0 = no pain 100 = worst pain imaginable
Pain score 10 hours post-operation | 10 hours postoperatively
  Visual analog scale pain scores 10 hours after the end of the operation.
  The visual analog scale is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The patient marks a point on the line that matches the amount of pain they feel.
  0 = no pain 100 = worst pain imaginable
Pain score 24 hours post-operation | 24 hours postoperatively
  Visual analog scale pain scores 24 hours after the end of the operation.
  The visual analog scale is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The patient marks a point on the line that matches the amount of pain they feel.
  0 = no pain 100 = worst pain imaginable
Pain score 48 hours post-operation | 48 hours postoperatively
  Visual analog scale pain scores 48 hours after the end of the operation.
  The visual analog scale is presented as a 100-mm horizontal line on which the patient's pain intensity is represented by a point between the extremes of "no pain at all" and "worst pain imaginable." The patient marks a point on the line that matches the amount of pain they feel.
  0 = no pain 100 = worst pain imaginable
Quality of Recovery Score 36 hours post-operation | 36 hours postoperatively
  Subjects will complete the 15-question Quality of Recovery 36 hours after the end of surgery. Scores will be compared to the baseline taken in the pre-operative hold area.
Quality of Recovery Score 48 hours post-operation | 48 hours postoperatively
  Subjects will complete the 15-question Quality of Recovery 48 hours after the end of surgery. Scores will be compared to the baseline taken in the pre-operative hold area.
Length of Stay | During hospitalization, approximately 5 days
  Length of stay in the hospital, defined as time between admission and discharge. Unit of measure: Days.
Incidence of nausea | During hospitalization, approximately 5 days
  A count of the incidences of treatment of nausea with medication.
Time to first flatus | 96 hours postoperatively
  Time of first flatus will be recorded by floor nurses and extracted from the electronic medical record. Unit of measure: Hours.
Time to first bowel movement | 96 hours postoperatively
  Time of first bowel movement will be recorded by floor nurses and extracted from the electronic medical record. Unit of measure: Hours.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Dominick, MD, Principal Investigator — Anesthesiologist; David Lunardini, MD, Principal Investigator — Orthopedic Surgeon
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hollmann MW, Durieux ME. Local anesthetics and the inflammatory response: a new therapeutic indication? Anesthesiology. 2000 Sep;93(3):858-75. doi: 10.1097/00000542-200009000-00038. No abstract available. PMID 10969322
- [Background] Marret E, Rolin M, Beaussier M, Bonnet F. Meta-analysis of intravenous lidocaine and postoperative recovery after abdominal surgery. Br J Surg. 2008 Nov;95(11):1331-8. doi: 10.1002/bjs.6375. PMID 18844267
- [Background] Martin F, Cherif K, Gentili ME, Enel D, Abe E, Alvarez JC, Mazoit JX, Chauvin M, Bouhassira D, Fletcher D. Lack of impact of intravenous lidocaine on analgesia, functional recovery, and nociceptive pain threshold after total hip arthroplasty. Anesthesiology. 2008 Jul;109(1):118-23. doi: 10.1097/ALN.0b013e31817b5a9b. PMID 18580181
- [Background] Farag E, Ghobrial M, Sessler DI, Dalton JE, Liu J, Lee JH, Zaky S, Benzel E, Bingaman W, Kurz A. Effect of perioperative intravenous lidocaine administration on pain, opioid consumption, and quality of life after complex spine surgery. Anesthesiology. 2013 Oct;119(4):932-40. doi: 10.1097/ALN.0b013e318297d4a5. PMID 23681143
- [Background] Kim KT, Cho DC, Sung JK, Kim YB, Kang H, Song KS, Choi GJ. Intraoperative systemic infusion of lidocaine reduces postoperative pain after lumbar surgery: a double-blinded, randomized, placebo-controlled clinical trial. Spine J. 2014 Aug 1;14(8):1559-66. doi: 10.1016/j.spinee.2013.09.031. Epub 2013 Nov 8. PMID 24216403